CLINICAL TRIAL: NCT01847612
Title: Evaluation of Indocyanine Green Fluorescent Cholangiography Versus Methylene Blue to Detect Postoperative Biliary Fistula After Hepatectomy: Randomized Controlled Study
Brief Title: Use of Indocyanine Green Cholangiography and Methylene Blue to Detect Postoperative Biliary Fistula After Hepatectomy
Acronym: CAMFIB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PI2013_843_0003; 2013-000408-40 (EudraCT Number)
Record Dates: First submitted 2013-04-30; First posted 2013-05-07 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Liver Disease
Keywords: per operative cholangiography; liver resection; biliary fistula
MeSH Terms: conditions — Liver Diseases; Biliary Fistula | interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- indocyanine green fluorescent cholangiography (Experimental): use of indocyanine green fluorescent cholangiography in the patients of this arm, an indocyanine green fluorescent cholangiography is performed
  Interventions: Procedure: indocyanine green fluorescent cholangiography
- methylene blue (Active Comparator): injection of methylene blue during the surgery
  Interventions: Drug: methylene blue

INTERVENTIONS:
Procedure: indocyanine green fluorescent cholangiography
  Arms: indocyanine green fluorescent cholangiography
Drug: methylene blue
  Arms: methylene blue

SUMMARY:
The aim of the present study is to evaluate whether the use of indocyanine green fluorescent cholangiography is responsible in a decrease of biliary fistula's rate in patients with liver diseases requiring liver resection.

ELIGIBILITY:
Inclusion Criteria:

* benin or malignant liver disease with resection of 2 or more segments
* liver resection by laparotomy
* written consent

Exclusion Criteria:

* previous hepatectomy
* emergency surgery
* allergy to indocyanine green
* allergy to methylene blue
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-07-08 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
biliary fistula rate | postoperative week 4
  the biliary fistula is defined as a bilirubin in the drain three times higher than the serum bilirubin.
  the primary endpoint will be evaluated by a medical committee composed by investigators not involved in the patients enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: jean marc regimbeau, MD, PhD, Principal Investigator — CHU amiens
Locations (1):
- Amiens University Hospital, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen-Khac E, Lobry C, Chatelain D, Fuks D, Joly JP, Brevet M, Tramier B, Mouly C, Hautefeuille V, Chauffert B, Regimbeau JM. A Reappraisal of Chemotherapy-Induced Liver Injury in Colorectal Liver Metastases before the Era of Antiangiogenics. Int J Hepatol. 2013;2013:314868. doi: 10.1155/2013/314868. Epub 2013 Mar 7. PMID 23533786